CLINICAL TRIAL: NCT06332209
Title: Addressing Barriers to Care Among Underserved Youth: Telehealth Delivery of Trauma-Focused Cognitive Behavioral Therapy - A Randomized Effectiveness-Implementation Trial
Brief Title: Randomized Trial of Tele Vs. Clinic TF-CBT in Puerto Rico
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Regan Stewart, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00135303; U66RH31458 (Other Grant/Funding Number: Telehealth Center of Excellence)
Record Dates: First submitted 2024-03-12; First posted 2024-03-27 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-01

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: trauma focused cognitive behavioral therapy; telehealth; community implementation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-TF-CBT (Active Comparator): Trauma-Focused Cognitive Behavioral Therapy delivered via telehealth
  Interventions: Behavioral: Trauma Focused Cognitive Behavioral Therapy
- Clinic-TF-CBT (Active Comparator): Trauma-Focused Cognitive Behavioral Therapy delivered in clinic (in-person)
  Interventions: Behavioral: Trauma Focused Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Trauma Focused Cognitive Behavioral Therapy — Trauma-Focused Cognitive-Behavioral Therapy (TF-CBT; Cohen et al., 2017) is an evidence-based, manualized treatment protocol designed to treat posttraumatic stress and co-occurring symptoms such as depression and anxiety in trauma-exposed children and youth and their supportive and non-offending caregivers. TF-CBT is divided into nine cognitive and behavioral components, all of which incorporate gradual exposure to trauma memories and reminders

SUMMARY:
The current study will evaluate TF-CBT delivered via tele-health for youth presenting with trauma symptoms via a randomized controlled trial. Goals of the current study are to examine the effectiveness of Tele-TF-CBT delivered by community providers in Puerto Rico in improving youth trauma outcomes. Goals are also to support the feasibility, acceptability, and engagement outcomes of Tele-health delivery.

DETAILED DESCRIPTION:
The current study will use a randomized controlled trial to examine telehealth delivery of Trauma Focused-Cognitive Behavioral Therapy (TF-CBT) for youth with trauma symptoms receiving care in community based clinics in Puerto Rico. First, the effectiveness of Tele-TF-CBT in improving trauma symptoms will be examined compared with clinic-based TF-CBT. Next, the feasibility, acceptability, and engagement outcomes of Tele-TF-CBT will be examined in this population. Lastly, implementation factors will be explored.

ELIGIBILITY:
Inclusion Criteria:

* 7-18 years old
* experienced at least one traumatic event
* present with clinically significant levels of post-traumatic stress symptoms

Exclusion Criteria:

* significant suicidal ideation
* substance use disorder
* active psychotic symptoms
* pervasive developmental delays,
* currently living with or in close contact with the perpetrator of their abuse

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Traumatic Stress Symptoms | baseline, post-treatment (2-weeks of completing treatment), 3-month follow-up (within 3 months of post-treatment assessment)
  Parent and youth rated trauma symptoms will be measured via the Child Post Traumatic Stress Disorder Symptoms Scale. Scores range from 0 to 80 with higher scores indicating higher levels of post traumatic stress.
Traumatic Stress Symptoms | baseline, post-treatment (2-weeks of completing treatment), 3-month follow-up (within 3 months of post-treatment assessment)
  Parent and youth rated trauma symptoms will be measured via the the UCLA Post Traumatic Stress Disorder Reaction Index Interview. Scores range from 0 to 80 with higher scores indicating higher levels of post traumatic stress.

SECONDARY OUTCOMES:
Anxiety and Depression Symptoms | baseline, post-treatment, 3-month follow-up
  Parent and youth rated anxiety and depression symptoms will be measured via the Revised Child Anxiety and Depression Scale Short form.Scores range from 0 to 75 with higher scores indicating higher levels of anxiety and depression.
Anxiety and Depression Symptoms | baseline, post-treatment (2-weeks of completing treatment), 3-month follow-up (within 3 months of post-treatment assessment)
  Parent and youth rated anxiety and depression symptoms will be measured via the Pediatric Symptom Checklist. Scores range from 0 to 70 with higher scores indicating higher levels of impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States